CLINICAL TRIAL: NCT00639834
Title: A Phase 1, Multicenter, Single-dose, Dose-escalation, Safety and Tolerability Study of MDX-1342 (Anti-CD19 Human Monoclonal Antibody) in Combination With Methotrexate in Subjects With Active Rheumatoid Arthritis
Brief Title: Study of the Safety of MDX-1342 in Combination With Methotrexate in Patients With Rheumatoid Arthritis
Acronym: MDX1342-01
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDX1342-01; IM130-001 (Other: BMS)
Record Dates: First submitted 2008-01-10; First posted 2008-03-20 (Estimated); Last update posted 2013-05-22 (Estimated); Status verified 2013-05

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid; arthritis; RA; joint inflammation; autoimmune; Medarex; Rheumatology
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis | interventions — MDX-1342 antibody

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Active MDX-1342 given in combination with Methotrexate
  Interventions: Biological: MDX-1342

INTERVENTIONS:
Biological: MDX-1342 — One dose of active MDX-1342 (anti-CD19 fully human monoclonal antibody) will be administered to patients as an i.v. infusion. Patients will receive one dose of MDX-1342 given in combination with Methotrexate treatment.

SUMMARY:
The purpose of this study is to determine if MDX-1342 given in combination with Methotrexate is a safe treatment for patients with active rheumatoid arthritis. In addition, changes in the severity patients' arthritis will also be analysed.

ELIGIBILITY:
Inclusion Criteria:

* Must have met ACR criteria for the diagnosis of rheumatoid arthritis (RA)
* Must have active RA
* Must be treated with Methotrexate (MTX) (10 to 25 mg weekly) for at least 3 months and have received a stable dose for at least 28 days prior to the anticipated study drug administration date.
* All other DMARDs or biologics must be discontinued at least 28 days prior to study drug administration and: 1) Leflunomide, which must be discontinued at least 60 days before study drug administration, 2) infliximab, adalimumab, and abatacept must be discontinued at least 56 days prior to study drug administration

Exclusion Criteria:

* Both Rheumatoid factor and anti-CCP negative
* Prior treatment with any B-cell depleting therapy
* Any other mAb or Ig-based fusion proteins 56 days or less prior to Visit
* History of or current inflammatory joint disease other than RA
* Neuropathies or neurovasculopathies that might interfere with pain evaluation
* Complications of RA or other disease
* Any other autoimmune disease other than RA
* Acute or chronic infection
* Clinically significant disease requiring

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2008-02; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
incidence and severity of treatment-emergent adverse events | all adverse events will be followed to resolution

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (24):
- United States (11):
  - Sun Valley Arthritis Center LTD., Peoria, Arizona
  - Impact Clinical Trials, Los Angeles, California
  - Centre for Rheumatology, Immunology and Arthritis (CRIA), Fort Lauderdale, Florida
  - Coastal Medical Research, Inc, Port Orange, Florida
  - Lovelace Scientific Resources, Venice, Florida
  - Good Samaritan Hospital and Johns Hopkins Hospital, Baltimore, Maryland
  - Justus Fiechtner, Lansing, Michigan
  - Columbia University Medical Center, New York, New York
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Arthritis Northwest Rheumatology, PLLC, Spokane, Washington
  - George Krick, MD, Tacoma, Washington
- Germany (3):
  - klinikum der Universitat zu Koln, Cologne
  - Universitatsklinikum "Carl Gustav Carus" an der Technischen Universtitat Dresden, Dresden
  - Klinikum rechts der Isar der TU Munchen, Munich
- Hungary (4):
  - DRC Gyógyszervizsgáló Központ Kft, Balatonfüred
  - Semmelweis Egyetem Altalanos Orvostudomanyi Kar-I. sz, Budapest
  - DEOEC Kinikai Farmakologiai Tanszek, Debrecen
  - First Department of Medicine, Szeged
- Ukraine (4):
  - V.K. Gusak Institute of Urgent & Reconstructive Surgery under UAMS, Hospital Therapy and Rehabilitaiton Clinic, Donetsk
  - Kharkiv Medical Academy of Postgraduate Education, City Clinical General Hospital #25, Kharkiv
  - Zaporizhya State Medical University, City Clinical Hopsital #6, Therapeutics Department, Zaporizhya
  - Zaporizhzhya Regional Clinical Hospital, Rheumatology Department, Zaporizhzhya
- United Kingdom (2):
  - The Kellgren Centre for Rheumatology, Manchester
  - Welcome Trust Clinical Research Facility, Southampton General Hospital, Southampton